CLINICAL TRIAL: NCT03472118
Title: Apneic Oxygenation Using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) in Adult Patients Undergoing Suspension Laryngoscopy Under General Anesthesia: a Multicenter Study
Brief Title: High Flow Oxygen in Patients Undergoing Suspension Laryngoscopy Under General Anesthesia
Acronym: OxALa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Risk-benefit analysis
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/04
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-03

CONDITIONS: Laryngoscopy; Apnea; Anesthesia
Keywords: Anesthesia, general; Adult; Humans; Apnea; Oxygen; Carbon dioxide; Acidosis, respiratory; Administration, Intranals/methods; Airway management/methods; Continuous positive airway pressure/methods; Insufflation/methods; Oxygen/administration&dosage; Laryngoscopy; Larynx/surgery
MeSH Terms: conditions — Apnea; Acidosis, Respiratory; Laryngeal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Flow Apneic Oxygenation (Experimental): Apneic oxygenation using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE)
  Interventions: Device: Nasal High Flow Oxygen

INTERVENTIONS:
Device: Nasal High Flow Oxygen — Nasal High Flow Oxygen during apnoea using Optiflow device of Fisher and Paykel

SUMMARY:
Patients undergoing suspension laryngoscopy under general anaesthesia have oxygen delivered to their lungs through different methods. Inserting a tube in the trachea is the best means for oxygen delivery. However, it does not allow for optimal visibility of the operated area. Other techniques can be used but have disadvantages with some being associated with serious complications. No consensus exists regarding the best airway management technique for this intervention.

The aim of the study is to investigate a new device that delivers oxygen at very high flow through a nasal cannula in patients undergoing suspension laryngoscopy under general anaesthesia. This technique allows the surgeon to have a perfect visualisation of the laryngeal structures while allowing the delivery of oxygen for the lungs.

After informed consent, adult patients undergoing suspension laryngoscopy under general anaesthesia in two French hospitals will receive high flow oxygen throughout the procedure. At the end of surgery or, whenever applicable, at the time of technique failure (with a decrease in blood oxygen saturation to less than 92%), blood will be drawn for analysis. All patients will have a thin security catheter inserted in their trachea (the currently used technique in both participating hospitals), allowing for rescue high frequency ventilation if ever the study technique fails.

The safety of the device will also be assessed by analysing the blood samples for signs of carbon dioxide accumulation and by collecting any intra or post-operative complications.

If the device shows to be effective at maintaining blood oxygenation without significant associated risks, it could be used for other surgical situations where airway management is expected to be difficult.

DETAILED DESCRIPTION:
Suspension laryngoscopy is a surgical intervention for which no airway management recommendations exist.

Many techniques are used, each having limitations. While tracheal intubation is the gold standard of airway management, in this particular intervention, it does not allow for optimal visualisation of the larynx. Maintaining spontaneous ventilation under general anaesthesia is used by some teams but puts the patient at the risk of laryngospasm. Apneic oxygenation is another option but its use is limited by the associated risk of hypercapnia. High frequency jet ventilation allows for good surgical conditions, satisfactory blood oxygen delivery and a low risk of hypercapnia; however, its use has been associated with severe, sometimes deadly, complications.

Nasal High Flow oxygenation is a relatively novel technique that allows for the delivery of heated and humidified oxygen with flow ranging up to 70l/min. It is widely used in neonatal and adult critical care. Its use in apneic patients under general anaesthesia has been reported to be associated with a mean of 14 minutes of desaturation-free apnea time with limited risk of hypercapnia. Desaturation-free apnea times up to 60 minutes have been reported. The use of nasal high flow apneic oxygenation in suspension laryngoscopy has been reported once in the literature with encouraging results.

The aim of the study is to assess the efficacy of nasal high flow oxygen in maintaining normal blood oxygen saturation (>95%) in apneic patients undergoing suspension laryngoscopy under general anaesthesia.

Adult patients undergoing suspension laryngoscopy (laser surgeries and cavoscopies excluded) in two french hospitals will be screened for eligibility by the anaesthesiologist during the preoperative consultation. Consenting and eligible patients will be enrolled in the study.

After pre oxygenation (until etO2 >90%), general anaesthesia will be started and maintained using TIVA propofol and remifentanil. Neuromuscular blockade will be achieved using rocuronium.

As soon as apnea is obtained, nasal high flow oxygen will be started at 70l/min using Simplified OptiflowTM (Fisher & Paykel Healthcare Ltd, Auckland, New Zealand) . A transglottic high frequency jet ventilation catheter will also be placed in the trachea to allow for emergency ventilation if high flow oxygenation fails to maintain SpO2>92%.

Oxygen saturation, blood pressure, pulse rate, BIS and neuromuscular blockade will be monitored throughout the surgery.

At the end of surgery (maximum 30 minutes), or as soon as blood oxygen saturation falls below 92%, whichever comes first, arterial blood for blood-gas analysis (PaO2, PaCO2, pH) will be drawn.

Neuromuscular blockade will be reversed with neostigmine or sugammadex depending on the depth of nerve block.

If the technique is shown to be associated with a low risk of blood oxygen desaturation and of severe hypercapnia, it could be considered for predictable difficult airway management.

ELIGIBILITY:
Inclusion Criteria:

* Consent for participation
* Affiliation to the french social security system
* Patients undergoing any suspension laryngoscopy other than laser surgery and cavoscopy and expected to last less than 30 minutes

Exclusion Criteria:

* Pregnancy
* Epilepsy
* Arrhythmia
* Pulmonary hypertension
* Lung disease with basal SpO2<95%
* Obstructive laryngeal tumor
* BMI>30kg.m-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence of oxygen desaturation SpO2<95% in the first fifteen minutes of apnea in patients undergoing suspension laryngoscopy under general anesthesia and receiving nasal high flow oxygen | throughout the first fifteen minutes following the start of apnea, ie following general anesthesia and neuromuscular blockade

SECONDARY OUTCOMES:
Incidence of oxygen desaturation SpO2<95% throughout surgery | throughout surgery (maximum thirty minutes)
Duration between start of apnea and oxygen desaturation spO2<95% | throughout surgery (maximum thirty minutes)
Incidence of hypercapnia (PaCO2>60mmHg) at the end of surgery or at technique failure | At the end of surgery (maximum thirty minutes) or at technique failure (upon blood oxygen desaturation SpO2<92%)

CONTACTS AND LOCATIONS:
Overall Officials: Mary SAAD, MD, Study Chair — Institut Curie
Locations (2):
- France (2):
  - Hôpital René Huguenin - Institut Curie, Saint-Cloud, Île-de-France Region
  - Hôpital Foch, Suresnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No